CLINICAL TRIAL: NCT06550973
Title: Randomized, Multicentric Trial, PROceeding With Advanced Techniques in Case of Distal Malignant Biliary Obstruction and Difficult Biliary Cannulation comparEd With Therapeutic-EUS: the PROMETHEUS Trial
Brief Title: PROceeding With Advanced Techniques in Case of Distal Malignant Biliary Obstruction and Difficult Biliary Cannulation comparEd With Therapeutic-EUS: the PROMETHEUS Trial
Acronym: PROMETHEUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4113
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Malignant Biliary Obstruction
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided biliary drainage (No Intervention): EUS-guided biliary drainage will be performed using a bi-flanged lumen apposing metal stent (LAMS) mounted on an electrocautery-enhanced delivery. After EUS identification of the dilated CBD, a place without interposing vessels will be found by the endosonographer. Transduodenal puncture of the CBD will be performed directly with the LAMS that will be used to cautery the tract and enter the CBD. The diameter and length of the stent and the modality of placing the stent (under complete EUS view or with endoscopic or fluoroscopic guidance) will be chosen at the discretion of the endoscopist performing the procedure.
- Rescue techniques (Experimental): Rescue techniques, such as pre-cut biliary sphincterotomy/fistulotomy, double guide wire (DGW) technique, wire-guided cannulation over a pancreatic stent and transpancreatic biliary sphincterotomy, will be used at the discretion of the endoscopist [12]. After deep cannulation, a cholangiogram to better define the characteristics of the stenosis will be done. The stent will then be inserted over a guidewire and deployed across the stenosis. All stents will be fully covered SEMSs or partially covered SEMSs of 10 mm diameter. The length of the stent will be chosen at the discretion of the endoscopist performing the procedure. A prophylactic pancreatic stent will be placed in patients who will be thought to be at high risk of post-procedure pancreatitis at the discretion of the treating endoscopist.
  Interventions: Procedure: pre-cut biliary sphincterotomy/fistulotomy, double guide wire (DGW) technique

INTERVENTIONS:
Procedure: pre-cut biliary sphincterotomy/fistulotomy, double guide wire (DGW) technique — Rescue techniques, such as pre-cut biliary sphincterotomy/fistulotomy, double guide wire (DGW) technique, wire-guided cannulation over a pancreatic stent and transpancreatic biliary sphincterotomy, will be used at the discretion of the endoscopist [12]. After deep cannulation, a cholangiogram to better define the characteristics of the stenosis will be done. The stent will then be inserted over a guidewire and deployed across the stenosis. All stents will be fully covered SEMSs or partially covered SEMSs of 10 mm diameter. The length of the stent will be chosen at the discretion of the endoscopist performing the procedure. A prophylactic pancreatic stent will be placed in patients who will be thought to be at high risk of post-procedure pancreatitis at the discretion of the treating endoscopist.
  Arms: Rescue techniques

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) stands as the primary approach for addressing jaundice in individuals with distal malignant biliary obstruction. A premise element in achieving success during therapeutic ERCP is selective biliary cannulation (SBC). Nevertheless, SBC doesn't consistently yield favorable outcomes, even among expert endoscopists, failing in around 25% to 50% of cases with standard ERCP approach (sphincterotome and guidewire).

In such situations, depending on the endoscopist's experience and preference, various advanced techniques come into play. These encompass the double guidewire cannulation approach, needle-knife precut papillotomy or fistulotomy, and transpancreatic sphincterotomy, serving as potential rescue methods.

In recent times, the EUS-guided approach has been gaining increasing significance. Initially, it was viewed as a rescue option in cases where advanced ERCP techniques failed (5-15% of cases). More recently, it has proved its feasibility as a first line alternative to ERCP in scenarios involving malignant biliary obstruction.

DETAILED DESCRIPTION:
Rationale of the study Patients with distal malignant biliary obstruction have a higher risk of ERCP failure, related to the difficulty of bile duct cannulation. These patients after standard ERCP strategies failure, undergo advanced ERCP rescue strategies and in case of failure to EUS guided biliary drainage. HoweverEUS guided biliary drainage performed following the attempted advanced ERCP strategies, it may carry the risk of adverse events of advance ERCP strategies. We hypothesize that, in this setting of patients, early EUS guided biliary drainage in case of difficult biliary cannulation has a lower risk of post-procedural adverse events, as well as better overall safety and efficacy profiles. This could imply better outcomes such as for those patients who are planned to receive a chemotherapy before surgery in which a complication, such as acute pancreatitis, could delay the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with distal malignant biliary obstruction
* Abdominal ultrasound or computed tomography or magnetic resonance or EUS showing a dilated common bile duct > 15 mm diameter.
* Difficult biliary cannulation defined as ESGE guidelines
* Agree to receive follow up phone calls
* Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders and/or INR>1.5, PLT<50,000 103/mm3.
* Use of anticoagulants that cannot be discontinued
* Pregnant women
* Previous ERCP or EUS-BD attempt
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of AE | 0 to 3 months
  such as the occurrence of unintentional perforation, bleeding requiring hemostasis, pancreatitis, stent malposition or migration, cholecystitis or cholangitis, jaundice, peritonitis, symptomatic bile leak, subcapsular liver hematoma, pneumoperitoneum, retained sheared wire, and procedure-related death

SECONDARY OUTCOMES:
Rate of any of the specific adverse events | 0 to 3 months
  such as the occurrence of unintentional perforation, bleeding requiring hemostasis, pancreatitis, stent malposition or migration, cholecystitis or cholangitis, jaundice, peritonitis, symptomatic bile leak, subcapsular liver hematoma, pneumoperitoneum, retained sheared wire, and procedure-related death
Rate of technical success | 0 to 3 months
  Defined as the rate of successful stent placement in the desired duct at the initial procedure)
Rate of clinical success | 0 to 3 months
  Defined as decrease of bilirubin level to either half the initial level, or less than 3 dl/mg -in order to allow to start chemotherapy
Time needed for technical success | during procedure
  duration of a successful procedure
Rate of reintervention | 0-3 months
  in the 3 months following the procedure, will evaluate the patients who need a reintervention
Rate of cross-over | 0-3 months
  Defined as in case of failure of the procedure established by the randomization the rate of crossover to the other procedure done.

IPD SHARING:
Plan to Share IPD: Undecided